CLINICAL TRIAL: NCT00067405
Title: Intravenous Micronutrient Therapy (IVMT) for Fibromyalgia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000942-01A1 (NIH); Katz
Record Dates: First submitted 2003-08-18; First posted 2003-08-20 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Intravenous micronutrient therapy; IVMT; alternative medicine; complementary medicine; vitamins; vitamin supplements
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Intravenous micronutrient therapy

SUMMARY:
The purpose of this study is to determine if intravenous micronutrient therapy (IVMT) is effective in the treatment of fibromyalgia, as assessed by validated functional and pain measures.

DETAILED DESCRIPTION:
As per Brief Summary

ELIGIBILITY:
Inclusion criteria:

* Meet the American College of Rheumatology criteria for Fibromyalgia diagnosis;
* On no medication for Fibromyalgia other than acetaminophen, or willing to stop all such medication for the duration of the study

  * Willing to stop all FMS medication for the duration of the study or be on a stable dose of such medication for at least 3 months

Exclusion criteria:

* Other concurrent medical conditions such as rheumatologic disease, chronic infection, untreated endocrine disorders, unstable seizures, psychiatric disorders, acute peptic ulcer disease, congestive heart failure, chronic liver disorders and/or bleeding problems

  * Allergy to thiamin
* Unwilling to stop vitamin supplementation for the duration of the study

  * PLEASE NOTE: Travel to and accomodations at the study site can NOT be compensated. Anyone wishing to travel from outside of the study site's geographic area must do so at their own risk and expense.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Katz, MD, Principal Investigator — Yale-Griffin Prevention Research Center
Locations (1):
- Yale-Griffin Prevention Research Center, Derby, Connecticut, United States

REFERENCES:
- [Derived] Ali A, Njike VY, Northrup V, Sabina AB, Williams AL, Liberti LS, Perlman AI, Adelson H, Katz DL. Intravenous micronutrient therapy (Myers' Cocktail) for fibromyalgia: a placebo-controlled pilot study. J Altern Complement Med. 2009 Mar;15(3):247-57. doi: 10.1089/acm.2008.0410. PMID 19250003